CLINICAL TRIAL: NCT05138523
Title: Observational, Open Label Study With Direct Individual Benefit Assessing the Efficacy and Safety of Sofosdac® 400mg/60mg Tablets (400 mg Sofosbuvir and 60 mg of Daclatasvir) Treatment in Patients With Chronic Hepatitis C (HCV)
Brief Title: Evaluation of the Efficacy and Safety of the Fixed-dose Combination Sofosdac® 400mg/60mg in Patients With Chronic Hepatitis C (HCV)
Status: Completed | Type: Observational
Sponsor: Beker Laboratories (Industry)
Collaborators: Pharmaceutical Research Unit, Jordan (Other)
Responsible Party: Sponsor
Other Study IDs: DASO2018/PRO-00
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Chronic Hepatitis c
Keywords: HCV; Cirrhotic; non-cirrhotic; sofosdac; sofosbuvir; daclatasvir; fixed-dose combination; FDC; hepatitis C; pangenotypic; genotype
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-cirrhotic: Non-cirrhotic HCV patients; 12 weeks treatment
  Interventions: Combination Product: Sofosdac®
- Cirrhotic: Cirrhotic HCV patients; 24 weeks treatment
  Interventions: Combination Product: Sofosdac®

INTERVENTIONS:
Combination Product: Sofosdac® — Once daily fixed-dose combination of 400 mg Sofosbuvir and 60 mg Daclatasvir

SUMMARY:
A multicentric, observational, open-design study conducted to evaluate the efficacy and safety of Sofosdac® 400mg/60mg tablets treatment in 100 patients with chronic hepatitis C (HCV)

DETAILED DESCRIPTION:
BEKER laboratories developed the generic drug Sofosdac® 400 mg/60 mg Tablets as fixed dose combination that contains two direct antiviral agents (400 mg Sofosbuvir and 60 mg Daclatasvir) known to be pangenotypic in order to fulfill WHO plan to eradicate HCV by 2030. BEKER conducted an observational clinical trial to evaluate the efficacy and safety of FDC Sofosdac® 400 mg/60 mg treatment in Algerian patients with chronic hepatitis C (HCV).

ELIGIBILITY:
Inclusion Criteria:

* Men and women age of 18 years old and older.
* HCV chronic Infection, genotype 1 or 2 or 3 or 4 or 5 or 6
* Naive
* Bi-therapy failure, Tri-therapy 1st generation Telaprévir and Boceprevir, Sofosbuvir - pegIFN - RBV failure
* Evaluation of fibrosis by non-invasive methods (Fibroscan, Fib 4, APRI) performed during the pre-inclusion period (of at least one month) or A Liver biopsy puncture of at least 24 months before the inclusion visit.
* Fibrosis according to Metavir score: F0, F1, F2, F3, F4.
* Compensated Cirrhosis Child-Pugh A or
* Decompensated Cirrhosis (This point is applicable for patients who have cirrhosis)

Exclusion Criteria:

* Patient under amiodarone
* Hepatocellular carcinoma HCC
* Haemodialysis
* Creatinine Clearance < 30ml/min
* Breastfeeding
* Impossibility of using effective masculine or feminine contraception during the study and 6 months after treatment cessation.
* Medications triggering conduction disturbances with long QT, 30 days prior to inclusion
* QT prolongation > 450 ms
* Personal or familial history of torsade de pointes
* Allergies to nucleosi(ti)des analogues.
* Advanced cardiopulmonary pathology
* Malignant neoplasia
* The intake of anticonvulsants: Carbamazepine, eslicarbazepine, fosphenytoin, phenytoin, oxcarbazepine, pentobarbital, phenobarbital, primidone or the antimycobacterial agents: Rifabutin, rifampin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in the study were enrolled from five centers (primary care facilities) across different regions in the country; East, Center and West of Algeria.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Detection of RNA HCV 12 weeks after treatment cessation by acceptable quantification assay | 12 weeks after treatment cessation
  A quantification assay is performed to all patients to detect RNA HCV in order to determine the proportion of patients who achieve SVR12 (Sustained Viral Response) defined as:
  RNA HCV < LLOQ (Lower Limit of Quantification) 12 weeks after treatment cessation.

SECONDARY OUTCOMES:
Assessment of reported adverse events | During treatment duration defined as: 24 weeks for cirrhotics, and 12 weeks for non-cirrhotic patients
  Assessment of observed adverse events / adverse effects and serious adverse events related or not related to Sofosdac® treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Debzi, MD; Professor, Principal Investigator — CHU Mustapha Hepatology department
Locations (4):
- Algeria (4):
  - Boufarik Public Hospital, Boufarik, Blida Province
  - Khenchla Public Hospital, Khenchla, Khenchla
  - Mustapha Pacha Teaching Hospital, Algiers
  - Oran Teaching Hospital, Oran

IPD SHARING:
Plan to Share IPD: Undecided
IPD collected will be available to other researchers upon their request.